CLINICAL TRIAL: NCT04692792
Title: Efficacy Evaluation of Dai Dai Flower on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH109-REC1-161
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Gastroenterology
Keywords: Obesity; Weight control; Dai Dai flower
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Dai Dai flower drink (Experimental)
  Interventions: Dietary Supplement: Dai Dai flower drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle (50 mL) per day for 8 weeks
  Arms: Placebo drink
Dietary Supplement: Dai Dai flower drink — consume 1 bottle (50 mL) per day for 8 weeks
  Arms: Dai Dai flower drink

SUMMARY:
To assess the Dai Dai flower extract on body weight control

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged between 20 and 60 years old
* Body mass index (BMI) ≥ 24 (kg/m^2) or body fat mass ≥ 25%

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Implementation in weight loss programs, consumption drugs or supplements for weight control before 3 months of this study
* Participate weight control or fat loss human studies before 3 months of this study
* History of cardiovascular disease, liver disease, kidney disease, endocrine disease, or other major organic diseases (according to subjects reporting).
* Person who has received major surgery or bariatric surgery (according to medical history).
* Person who has received constant drug use.
* People with mental illness

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The change of body weight | Change from Baseline body weight at 8 weeks
  The body weight (kg) was assessed by InBody.
The change of BMI | Change from Baseline BMI at 8 weeks
  The BMI was assessed by InBody.

SECONDARY OUTCOMES:
The change of body fat mass | Change from Baseline body fat mass at 8 weeks
  The body fat mass (kg) was assessed by InBody.
The change of visceral fat mass | Change from Baseline visceral fat mass at 8 weeks
  The visceral fat mass (kg) was assessed by InBody.
The change of waist-hip ratio | Change from Baseline waist-hip ratio at 8 weeks
  The waist-hip ratio was assessed by measuring tape.
The change of basal metabolic rate | Change from Baseline basal metabolic rate at 8 weeks
  The basal metabolic rate was assessed by InBody.
The change of AST | Change from Baseline AST at 8 weeks
  Venous blood was sampled to measure concentrations of aspartate transaminase (AST)
The change of ALT | Change from Baseline ALT at 8 weeks
  Venous blood was sampled to measure concentrations of alanine aminotransferase (ALT)
The change of Creatinine | Change from Baseline creatinine at 8 weeks
  Venous blood was sampled to measure concentrations of creatinine
The change of BUN | Change from Baseline BUN at 8 weeks
  Venous blood was sampled to measure concentrations of blood urea nitrogen (BUN)
The change of fasting glycemia | Change from Baseline fasting glycemia at 8 weeks
  Venous blood was sampled to measure concentrations of fasting glycemia
The change of total cholesterol | Change from Baseline total cholesterol at 8 weeks
  Venous blood was sampled to measure concentrations of total cholesterol
The change of triglyceride | Change from Baseline triglyceride at 8 weeks
  Venous blood was sampled to measure concentrations of triglyceride
The change of HDL-cholesterol | Change from Baseline HDL-cholesterol at 8 weeks
  Venous blood was sampled to measure concentrations of HDL-cholesterol
The change of LDL-cholesterol | Change from Baseline LDL-cholesterol at 8 weeks
  Venous blood was sampled to measure concentrations of LDL-cholesterol
The change of insulin | Change from Baseline insulin at 8 weeks
  Venous blood was sampled to measure concentrations of insulin
The change of adiponectin | Change from Baseline adiponectin at 8 weeks
  Venous blood was sampled to measure concentrations of adiponectin
The change of leptin | Change from Baseline leptin at 8 weeks
  Venous blood was sampled to measure concentrations of leptin
The change of IFN-γ | Change from Baseline IFN-γ at 8 weeks
  Venous blood was sampled to measure concentrations of IFN-γ
The change of IL-2 | Change from Baseline IL-2 at 8 weeks
  Venous blood was sampled to measure concentrations of IL-2
The change of IL-1beta | Change from Baseline IL-1beta at 8 weeks
  Venous blood was sampled to measure concentrations of IL-1beta

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Mei Chiang, Prof., Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan